CLINICAL TRIAL: NCT00899977
Title: A Double-blind, Randomized, Placebo-controlled, Sequential Group Pilot Study to Assess Safety, Tolerability, and Effectiveness of TC-5214 as Augmentation Therapy in Patients With Refractory Hypertension
Brief Title: TC-5214 as Augmentation Therapy in Patients With Refractory Hypertension
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TC-5214-23-CRD-002
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Refractory Hypertension
Keywords: refractory hypertension; hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Subjects may receive a single, oral dose of placebo (capsule) in one of 4 crossover periods. Also, subjects may receive placebo orally, twice daily for 14 days in the last phase of the study.
  Interventions: Drug: Placebo
- 1 mg TC-5214 (Experimental): Subjects may receive a single, oral capsule of 1 mg TC-5214 in one of 4 crossover periods.
  Interventions: Drug: TC-5214
- 2 mg TC-5214 (Experimental): Subjects may receive a single, oral capsule of 2 mg TC-5214 in one of 4 crossover periods.
  Interventions: Drug: TC-5214
- 4 mg TC-5214 (Experimental): Subjects may receive a single, oral capsule of 4 mg TC-5214 in one of 4 crossover periods. Also, subjects may receive 4 mg TC-5214 orally, twice daily for 14 days in the last phase of the study.
  Interventions: Drug: TC-5214
- 8 mg TC-5214 (Experimental): Subjects may receive a single, oral capsule of 8 mg TC-5214 in one of 4 crossover periods.
  Interventions: Drug: TC-5214

INTERVENTIONS:
Drug: Placebo — Matching placebo
  Arms: Placebo
Drug: TC-5214
  Arms: 1 mg TC-5214; 2 mg TC-5214; 4 mg TC-5214; 8 mg TC-5214

SUMMARY:
A pilot study of subjects with refractory hypertension (on 3 concomitant agents with SBP > 140 mmHg and a DBP > 90 mmHg) randomized in a double-blind fashion to receive 4 single escalating doses of study medication in clinic.

DETAILED DESCRIPTION:
12 subjects with refractory hypertension will be randomized in a double-blind fashion to receive single escalating doses of study medication in-clinic: on Day 1 (1mg), Day 8 (2mg), Day 15 (4mg) and Day 22 (8mg). On each of these 4 days, 10 subjects will receive TC-5214, and 2 subjects will receive placebo. Placebo treatments will be pooled across the 4 days of single-dose to produce an equivalent reference cohort (n = 8) for each treatment dose (n=10). Following the single-dose administration of 8mg in the clinic on Day 22, subjects will continue with two weeks (Days 23 - 35) of outpatient self-administration of TC-5214 (4mg BID; n = 6), or matching placebo (BID; n = 6). On Day 36, subjects will return for a final in-clinic dose of either TC-5214 (4mg, n = 6) or placebo (n = 6). There will be a 1-week follow-up period at the end of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory hypertension, defined as a SBP of >140mmHg and a DBP > 90mmHg, on stable doses of at least 3 concomitant antihypertensive treatment (which must include a diuretic and an ACEI, ARB or RA) for 8 weeks prior to Screening. All approved antihypertensive treatments are allowed except for alpha-adrenergic blockers, hydralazine, clonidine, guanethidine, guanadrel, and rauwolfia alkaloids.
2. Stable hypertension, as defined by: a. mean SBP on Day -7 that is within 20mmHg of the mean SBP on Day 1, with both mean SBPs > 140mmHg; and b. mean DBP on Day -7 that is within 10mm of the mean DBP on Day 1, with both mean DBPs > 90mmHg.
3. Outpatient with stable housing.
4. Subjects must be able to stay in the clinic for 8 hrs on Day 1, Day 8, Day 15, Day 22, and Day 36.
5. Able to give and to sign informed consent.

Exclusion Criteria:

1. Any unstable medical condition other than hypertension;
2. Stage 3 hypertension (SBP > 180mmHg and/or DBP > 110mmHg);
3. Heart rate > 100 beats per minute;
4. WOCBP who is pregnant or who is planning to become pregnant during the study;
5. History within past year of alcohol or illicit drug abuse;
6. Unable to comply with study procedures in opinion of investigator;
7. Concomitant medications for any medical condition that is uncontrolled for more than 2 weeks prior to study entry;
8. Current use of alpha-adrenergic blocker, hydralazine, clonidine, guanethidine, guanadrel, or rauwolfia alkaloids;
9. History of myocardial infarction or angina pectoris;
10. Current seizure disorder;
11. Renal insufficiency as defined by a serum creatinine > 2.0;
12. Uncontrolled hypothyroidism, vitamin B12 or folic acid deficiency;
13. History of or concurrent ileus, glaucoma, or urinary retention;
14. Inability of subject to understand and sign the ICF;
15. Known systemic infection (HBV, HCV, HIV, TB);
16. Current use of smoking cessation therapy within 4 weeks of screening;
17. Use of herbal supplements;
18. Clinically significant finding on physical exam;
19. Clinically significant laboratory or ECG abnormality, including QTcF > 460 msec;
20. Participation in another clinical trial in last month;
21. Body Mass Index (BMI) > 35.
22. Body weight < 100 pounds.
23. Site staff or family member of study site staff.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Mean difference between TC-5214 and placebo in change at 3 hours from baseline SBP | Following dosing, 3 manual seated BP measurements and orthostatic BP measurements will be obtained in an identical fashion, at 30 minutes post-dose and at 1, 2, 3, 4, 5, 6, 7, and 8 hrs post-dose.

SECONDARY OUTCOMES:
Safety and tolerability of TC-5214 in patients with refractory hypertension and obtain preliminary dose-response estimates | Days 1, 8, 15, 22 and 36

CONTACTS AND LOCATIONS:
Locations (1):
- Piedmont Medical Research, Winston-Salem, North Carolina, United States